CLINICAL TRIAL: NCT06404515
Title: Utilizing Telehealth Group Counseling Sessions to Improve the Process and Delivery of Secondary Preventive Care for Women With Atherosclerotic Cardiovascular Disease
Brief Title: Telehealth Group Counseling and Preventive Care for Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-03023409
Record Dates: First submitted 2024-04-30; First posted 2024-05-08 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: ASCVD; NSTEMI; STEMI; Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction; Unstable Angina; Chest Pain
Keywords: ASCVD; NSTEMI; STEMI; Coronary Artery Disease; ACS; Myocardial Infarction; Unstable Angina; Chest Pain
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction; Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable; Chest Pain

STUDY DESIGN:
Intervention Model Description: Subjects will participate in at least one telehealth session, lasting one hour, or up to five sessions lasting one hour each, over the course of 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth Counseling (Experimental): Telehealth sessions
  Interventions: Other: Telehealth Group Counseling

INTERVENTIONS:
Other: Telehealth Group Counseling — Group counseling for women via telehealth to provide educational materials about atherosclerotic heart disease and provide information about risk factors and modification of risk factors. Women then have an opportunity to discuss / ask questions.

SUMMARY:
The purpose of this study is to utilize an innovative healthcare delivery strategy via telehealth group counseling sessions to improve engagement, adherence, and ultimately outcomes in female patients with atherosclerotic cardiovascular disease (ASCVD).

DETAILED DESCRIPTION:
This will be an electronic survey study of female patients with known atherosclerotic cardiovascular disease (ASCVD) who are managed by providers in the Weill Cornell Medicine Cardiology Division and self-select into this telehealth group education series. Group health counseling will be administered via the Weill Cornell Medicine approved telehealth platform at the time of participation. Participants will have the option to choose the session topic of their choice and will have the opportunity to participate in 1-5 sessions over 12 weeks, depending on their preference. Each session will occur regardless of number of participants but will be capped at 12 participants, anticipating that two will not join. Once consent is obtained, baseline characteristics of participants will be collected via chart review. Demographics such as age, race, insurance carrier, and clinician-documented diagnoses, such as ASCVD, hypertension (HTN), hyperlipidemia (HLD), and diabetes mellitus (DM), will be collected. Prior to each group health counseling session, an initial survey will be provided to patients who are chosen for and consent to this study. This survey will ask patients about their demographics, self-reported diagnoses, current level of satisfaction about their understanding of their diagnoses, reasons for participating in the study, and history of previous participation in telehealth group counseling. After the sessions, a post-session survey will be provided to all participants and will assess patient understanding, including diagnoses and medications, satisfaction with the format, satisfaction with the provider, how many sessions were attended, reasons for attending more than one session, and recommendation of this format to others. All data will be de-identified prior to analysis and will remain confidential among investigators.

ELIGIBILITY:
Inclusion criteria:

* Female patients
* Age 18 and older
* Patients who are managed by providers at the Weill Cornell Medicine Women's Heart Program
* Women with evidence of atherosclerotic cardiovascular disease (ASCVD) and diagnoses of chest pain, myocardial infarction/heart attack (myocardial infarction - non ST elevation NSTEMI, ST elevation STEMI), coronary artery disease, acute coronary syndrome, unstable angina, atherosclerotic cardiovascular disease, hypertension (HTN), hyperlipidemia (HLD), diabetes (DM), and/or palpitations (as confirmed by clinician referral to study and chart review)

Exclusion criteria:

• Women with risk factors (ex: HTN, HLD, DM) but no evidence of ASCVD

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Change in patient's accessibility to care as assessed by Likert scale. | Immediately Before and Immediately After Each Counseling Session, up to 12 weeks
  Score ranges from 0 to 5 with 0 being not satisfied and 5 being very satisfied.
Change in patient's understanding of their disease as assessed by Likert scale. | Immediately Before and Immediately After Each Counseling Session, up to 12 weeks
  Score ranges from 0 to 5 with 0 being not satisfied and 5 being very satisfied.
Change in medication compliance as assessed by Likert scale. | Immediately Before and Immediately After Each Counseling Session, up to 12 weeks
  Score ranges from 0 to 5 with 0 being not likely and 5 being very likely.
Change in overall patient satisfaction as assessed by Likert scale. | Immediately Before and Immediately After Each Counseling Session, up to 12 weeks
  Score ranges from 0 to 5 with 0 being not satisfied and 5 being very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Diala Steitieh, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aggarwal NR, Patel HN, Mehta LS, Sanghani RM, Lundberg GP, Lewis SJ, Mendelson MA, Wood MJ, Volgman AS, Mieres JH. Sex Differences in Ischemic Heart Disease: Advances, Obstacles, and Next Steps. Circ Cardiovasc Qual Outcomes. 2018 Feb;11(2):e004437. doi: 10.1161/CIRCOUTCOMES.117.004437. PMID 29449443
- [Background] Mosca L, Barrett-Connor E, Wenger NK. Sex/gender differences in cardiovascular disease prevention: what a difference a decade makes. Circulation. 2011 Nov 8;124(19):2145-54. doi: 10.1161/CIRCULATIONAHA.110.968792. PMID 22064958
- [Background] Okunrintemi V, Valero-Elizondo J, Patrick B, Salami J, Tibuakuu M, Ahmad S, Ogunmoroti O, Mahajan S, Khan SU, Gulati M, Nasir K, Michos ED. Gender Differences in Patient-Reported Outcomes Among Adults With Atherosclerotic Cardiovascular Disease. J Am Heart Assoc. 2018 Dec 18;7(24):e010498. doi: 10.1161/JAHA.118.010498. PMID 30561253
- [Background] Garcia M, Mulvagh SL, Merz CN, Buring JE, Manson JE. Cardiovascular Disease in Women: Clinical Perspectives. Circ Res. 2016 Apr 15;118(8):1273-93. doi: 10.1161/CIRCRESAHA.116.307547. PMID 27081110
- [Background] Fiscella K, Epstein RM. So much to do, so little time: care for the socially disadvantaged and the 15-minute visit. Arch Intern Med. 2008 Sep 22;168(17):1843-52. doi: 10.1001/archinte.168.17.1843. PMID 18809810
- [Background] Tai-Seale M, McGuire TG, Zhang W. Time allocation in primary care office visits. Health Serv Res. 2007 Oct;42(5):1871-94. doi: 10.1111/j.1475-6773.2006.00689.x. PMID 17850524
- [Background] Duryee R. The efficacy of inpatient education after myocardial infarction. Heart Lung. 1992 May;21(3):217-25. PMID 1592611
- [Background] Theis SL, Johnson JH. Strategies for teaching patients: a meta-analysis. Clin Nurse Spec. 1995 Mar;9(2):100-5, 120. doi: 10.1097/00002800-199503000-00010. PMID 7600475
- [Background] Winslow E, Bohannon N, Brunton SA, Mayhew HE. Lifestyle modification: weight control, exercise, and smoking cessation. Am J Med. 1996 Oct 8;101(4A):4A25S-31S; discussion 31S-33S. doi: 10.1016/s0002-9343(96)00317-8. PMID 8900334
- [Background] Kingsbury K. Taking AIM: how to teach primary and secondary prevention effectively. Can J Cardiol. 1998 Apr;14 Suppl A:22A-26A. PMID 9594930
- [Background] US Preventive Services Task Force; Grossman DC, Bibbins-Domingo K, Curry SJ, Barry MJ, Davidson KW, Doubeni CA, Epling JW Jr, Kemper AR, Krist AH, Kurth AE, Landefeld CS, Mangione CM, Phipps MG, Silverstein M, Simon MA, Tseng CW. Behavioral Counseling to Promote a Healthful Diet and Physical Activity for Cardiovascular Disease Prevention in Adults Without Cardiovascular Risk Factors: US Preventive Services Task Force Recommendation Statement. JAMA. 2017 Jul 11;318(2):167-174. doi: 10.1001/jama.2017.7171. PMID 28697260
- [Background] Manocchia A. Telehealth: Enhancing Care through Technology. R I Med J (2013). 2020 Feb 3;103(1):18-20. PMID 32013298